CLINICAL TRIAL: NCT05337176
Title: Impact of Sleeve Gastrectomy on Balance and Cognitive Function: A Cross-sectional Study
Brief Title: Impact of Sleeve Gastrectomy on Balance and Cognitive Function
Status: Completed | Type: Observational
Sponsor: Rawan Alwafi (Other)
Responsible Party: Sponsor-Investigator, Rawan Alwafi, Impact of Sleeve Gastrectomy on Balance and Cognitive Function: A Cross-sectional study, Umm Al-Qura University
Organization: Umm Al-Qura University (Other)
Other Study IDs: UmmAlQura
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Effect of Sleeve Gastrostomy in Both Cognition and Balance
Keywords: sleeve gastrectomy; Balance; cognition
MeSH Terms: interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: app-coo application — The Montreal Cognitive Assessment (MoCA) is a measure designed specifically for detecting mental cognitive impairment(MCI) APP-Coo-Balance-Test can assess the oscillation of the trunk in different static positions: "Feet Together", "On a Broad Base" (medial malleoli 30 cm apart) , and during the gait "Dynamic"(Arcuria et al., 2020).
  Other Names: MoCA (Montreal cognitive assessment)

SUMMARY:
Purpose of the study:

Purpose of study is to determine the effect of sleeve gastrectomy on balance and cognitive function in Saudi Arabia.

Aim of study:

To investigate if there is any change of balance and cognitive function disturbance after sleeve gastrectomy on participant.

Research hypothesis:

Sleeve gastrectomy have no impact on balance and cognitive function.

Inclusion criteria:

The participant will be selected according to the following criteria: 1.History of sleeve gastrectomy within 1 to 5 years.

2. Their age between (20-60 years). 3.Ability to walk without any assistive device. 4.All participant should be able to understand all requested instructions

Exclusion criteria:

The participant will be excluded if they have:

1. Any cognitive disturbances.
2. Disease that may affect balance (Spinal stenosis, peripheral polyneuropathy, vestibular impairment).
3. Gastrectomy operation less than 1year.
4. Pregnancy.

Material:

1. Introduction survey (willingness of participant) to recruit sittable participant.
2. Assessment form survey to collected data and result (include MOCA and App-coo application)

ELIGIBILITY:
Inclusion Criteria:

-

The participant will be selected according to the following criteria:

1. History of sleeve gastrectomy within 1 to 5 years.
2. Their age between (20-60 years).
3. Ability to walk without any assistive device.
4. All participant should be able to understand all requested instructions

Exclusion Criteria:

-

The participant will be excluded if they have:

1. Any cognitive disturbances.
2. Disease that may affect balance (Spinal stenosis, peripheral polyneuropathy, vestibular impairment).
3. Gastrectomy operation less than 1year.

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: participants for gender (male and Female) , age ranged from 20 to 60 years old, were randomly involved After bariatric surgery from different regions across Saudi Arabia
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
impact of sleeve gastrectomy on cognition | 2 to 3 month
  by using (MoCA) and see the result

SECONDARY OUTCOMES:
impact of sleeve gastrectomy on balance | 2 to 3 months
  by using a new application called : app-coo balance test

CONTACTS AND LOCATIONS:
Locations (1):
- Rawan Alwafi, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No